CLINICAL TRIAL: NCT00062764
Title: Long-Term Treatment of Nonalcoholic Steatohepatitis With Pioglitazone
Brief Title: Treating Nonalcoholic Steatohepatitis With Pioglitazone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jay Hoofnagle, Principal Investigator, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030212; 03-DK-0212
Record Dates: First submitted 2003-06-12; First posted 2003-06-13 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis
Keywords: Insulin Resistance; Obesity; Fatty Liver; Cirrhosis; Diabetes; Pioglitazone; Thiazolidinediones; Peroxisome Proliferator-Advanced Receptor Gamma; PPAR Gama; Nonalcoholic Steatohepatitis; Hepatitis; Non-Alcoholic Steatohepatitis; NASH
MeSH Terms: conditions — Hepatitis; Insulin Resistance; Obesity; Fatty Liver; Fibrosis; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental)
  Interventions: Drug: Actos (Pioglitazone)

INTERVENTIONS:
Drug: Actos (Pioglitazone) — Pts receive drug in a dose of 15 mg daily for at least 1 year; the dose is escalated to 30 mg daily if serum ALT levels do not fall to normal by the 1 year pt; if pts have a biochemical response, drug is continued for 3 years,

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is a common liver disease that resembles alcoholic hepatitis but occurs in persons who drink little or no alcohol. The etiology of NASH is unclear, but it is commonly associated with diabetes, obesity, and insulin resistance. Several pilot studies, including a study of pioglitazone at the NIH Clinical Center (01-DK-0130), have shown that the insulin-sensitizing thiazolidinediones lead to decreases in serum alanine aminotransferase (ALT) levels and improved liver histology. Once therapy is stopped, however, ALT levels rapidly return to pre-treatment values. Inaddition we are currently enrolling patients with NASH in a pilot study of metformin therapy for 48-weeks, however our results in 3 patients thus far have not been very encouraging.

In the current study, patients who have completed the pilot study of pioglitazone and have been off therapy for 48 weeks will be offered re-treatment for 3 years. We also propose to treat patients who have not had a satisfactory response to metformin with pioglitazone for the same duration. After a repeat medical and metabolic evaluation and liver biopsy, patients with moderate-to-severe NASH (activity score greater than or equal to 4) will restart pioglitazone at a dose of 15 mg daily. If after 48 weeks, ALT levels are not normal or improved to the degree identified during the pilot study, the dose will be increased to 30 mg daily at the end of 3 years, all patients will undergo repeat medical and metabolic evaluation and liver biopsy. The primary end point will be improvement in liver histology. Secondary end points will be improvements in insulin sensitivity, reduction in visceral fat, liver volume, and liver biochemistry. The aim of this study is to evaluate whether long-term pioglitazone therapy can safely achieve and maintain biochemical and histological improvements in NASH.

...

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis (NASH) is a common liver disease that resembles alcoholic hepatitis but occurs in persons who drink little or no alcohol. The etiology of NASH is unclear, but it is commonly associated with diabetes, obesity, and insulin resistance. Several pilot studies, including a study of pioglitazone at the NIH Clinical Center (01-DK-0130), have shown that the insulin-sensitizing thiazolidinediones lead to decreases in serum alanine aminotransferase (ALT) levels and improved liver histology. Once therapy is stopped, however, ALT levels rapidly return to pre-treatment values. Inaddition we are currently enrolling patients with NASH in a pilot study of metformin therapy for 48-weeks, however our results in 3 patients thus far have not been very encouraging.

In the current study, patients who have completed the pilot study of pioglitazone and have been off therapy for 48 weeks will be offered re-treatment for 3 years. We also propose to treat patients who have not had a satisfactory response to metformin with pioglitazone for the same duration. After a repeat medical and metabolic evaluation and liver biopsy, patients with moderate-to-severe NASH (activity score greater than or equal to 4) will restart pioglitazone at a dose of 15 mg daily. If after 48 weeks, ALT levels are not normal or improved to the degree identified during the pilot study, the dose will be increased to 30 mg daily at the end of 3 years, all patients will undergo repeat medical and metabolic evaluation and liver biopsy. The primary end point will be improvement in liver histology. Secondary end points will be improvements in insulin sensitivity, reduction in visceral fat, liver volume, and liver biochemistry. The aim of this study is to evaluate whether long-term pioglitazone therapy can safely achieve and maintain biochemical and histological improvements in NASH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Completion of a 48-week course of pioglitazone in protocol 01-DK-0130 or completion of 48-weeks of metformin in protocol 03-DK-0233.

At least 48 weeks of follow up on no thiazolidinedione therapy after completion of protocol 01-DK-0130.

At least 24-weeks follow up on no metformin theray after completion of protocol 03-DK-0233.

Written informed consent.

Patients who participated in protocol 01-DK-0130 will also have to meet the following inclusion criteria:

Demonstrated improvements in liver histology and/or serum ALT levels during the 48-week course of pioglitazone therapy in protocol 01-DK-0130.

Elevations in serum ALT levels.

Liver biopsy showing NASH with a total NASH activity score of at least 4 (of a total possible score of 16) including a score of at least 1 each for parenchyma inflammation, cellular injury and steatosis on liver biopsy taken 48 weeks after stopping pioglitazone.

Willingness to receive pioglitazone for 3 years.

Patients who participated in protocol 03-DK-0233 will also have to me the following inclusion criteria:

Demonstrated no significant improvement in liver histology and/or serum ALT levels during the 48-week course of metformin treatment in protocol 03-DK-0233.

Elevations in serum ALT levels.

Liver biopsy showing NASH with a total activity score of at least 4 (of a total possible score of 16) including a score of at least 1 each for parenchymal inflammation, cellular injury and steatosis on liver biopsy taken at the end of the 48-week course of metofrmin.

EXCLUSION CRITERIA:

Evidence of another form of liver disease (these largely will have been excluded based upon enrollment in the previous study, 01-DK-0130 and 03-DK-0233).

Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).

Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA in serum.

Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.

Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.

e. Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.

Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.

Hemochromatosis as defined by presence of 3+ or 4 iron on liver biopsy stain and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.

Drug-induced liver disease as defined on the basis of typical exposure and history.

Bile duct obstruction as shown by imaging studies.

History of excess alcohol ingestion, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1 drink per day: 7 drinks per week) in the previous one year.

Contraindications to liver biopsy: platelet counts less than 75,000/mm(3) or prothrombin time greater than 16 seconds.

Decompensated liver disease, Child-Pugh score greater than or equal to 7 points.

History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.

Preexistent diabetes mellitus or the development of diabetes mellitus during the study requiring the use of another drug in addition to pioglitazone for glycaemic control. Diabetes being as defined by: fasting plasma glucose of greater than or equal to 126 mg/dl on two separate occasions, or diabetic symptoms with a random plasma glucose of greater than or equal to 200 mg/dl.

Use of anti-diabetic drugs, including insulin, biguanides, sulfonylureas, or thiazolidinediones at the time of enrollment or in the previous 48 weeks.

Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator would preclude treatment with pioglitazone and adequate follow up.

Positive test for anti-HIV.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.

Pregnancy or inability to practice adequate contraception in women of childbearing potential.

Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study that is suggestive of liver cancer.

Any other conditions, which, in the opinion of the investigators would impede competence or compliance or possibility, hinder completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hoofnagle, MD, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Byron D, Minuk GY. Clinical hepatology: profile of an urban, hospital-based practice. Hepatology. 1996 Oct;24(4):813-5. doi: 10.1002/hep.510240410. PMID 8855181
- [Background] Ludwig J, Viggiano TR, McGill DB, Oh BJ. Nonalcoholic steatohepatitis: Mayo Clinic experiences with a hitherto unnamed disease. Mayo Clin Proc. 1980 Jul;55(7):434-8. PMID 7382552
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2001 and April 2002, 25 patients suspected of having NASH were evaluated, and 18 were enrolled in the study after screening.
Groups:
- Pioglitazone: Patients receive Pioglitazone in a dose of 15 mg daily for at least 1 year; the dose is escalated to 30 mg daily if serum Alanine transaminase levels do not fall to normal by the 1 year pt; if patients have a biochemical response, drug is continued for 3 years.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 3
  White | 13
  Mixed | 2
Region of Enrollment [Number; unit: participants]
  United States | 18
Obesity Distribution [Number; unit: participants]
  BMI>30 | 11
  BMI<=30 | 7
2-hr glucose diabetes mellitus [Number; unit: participants]
  >200 mg/dL | 2
  <=200 mg/dL | 16
2-hr glucose (Impaired glucose tolerance) [Number; unit: participants]
  140-199 mg/dL | 11
  other | 7
Metabolic syndrome [Number; unit: participants]
  Yes | 7
  No | 11
Fasting glucose [Number; unit: participant]
  110-125 mg/dL | 2
  other | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improvement in Liver Histology
Description: A histological response was defined as a reduction in the NASH activity index by 3 points or more with improvements of at least 1 point each in steatosis, parenchymal inflammation, and hepatocellular injury.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
participants | 12

2. Secondary Outcome: Number of Patients With Impaired Glucose Tolerance After Treatment
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
participants | 6

3. Secondary Outcome: Mean Increase of Insulin Sensitivity Index
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
percentage | 126 (78)

4. Secondary Outcome: Average Increase in Weight After Treatment
Time Frame: 48 weeks
Measure: Mean (Full Range); unit: kg
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
kg | 3.5 [-1.7 to 13.3]

5. Secondary Outcome: Mean BMI Change
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Pioglitazone
Number analyzed (Participants) | 18
kg/m2 | 1.3 (1.7)
Statistical Analysis 1: Comparison: Pioglitazone; Test type: Superiority or Other; p = 0.004, paired t-test

ADVERSE EVENTS:
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=18)
Worsened serum ALT levels (Gastrointestinal disorders) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=18)
dizziness (General disorders) | 1 (1)
Weight gain (General disorders) | 13 (13)

LIMITATIONS AND CAVEATS:
A major limitation of this study was the lack of a concurrently followed control group.

Another important shortcoming of this study was that patients were treated for 48 weeks only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes